CLINICAL TRIAL: NCT02307851
Title: A Phase 2 Randomized, Observer-Blind, Dose-Ranging Study to Evaluate the Immunogenicity and SAfety of Quadrivalent Seasonal Virus-Like Particle (VLP) Influenza Vaccine (Recombinant) in Healthy Young (18-49) Adults
Brief Title: Quadrivalent Influenza VLP Vaccine Dose Ranging Study in Young Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novavax (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FLU-SIQ-206
Record Dates: First submitted 2014-11-17; First posted 2014-12-04 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Experimental): Quadrivalent VLP vaccine, low dose, intramuscular injection (0.5mL)
  Interventions: Biological: Quadrivalent VLP Vaccine
- Group B (Experimental): Quadrivalent VLP vaccine, high dose, intramuscular injection (0.5mL)
  Interventions: Biological: Quadrivalent VLP Vaccine
- Group C (Experimental): Quadrivalent VLP vaccine, medium dose, intramuscular injection (0.5mL)
  Interventions: Biological: Quadrivalent VLP Vaccine
- Group D (Active Comparator): Comparator TIV, intramuscular injection (0.5mL)
  Interventions: Biological: Comparator TIV

INTERVENTIONS:
Biological: Quadrivalent VLP Vaccine
  Arms: Group A; Group B; Group C
Biological: Comparator TIV
  Arms: Group D

SUMMARY:
The purpose of this study is to determine the immune response of three dose levels of the Quadrivalent VLP vaccine in healthy young (18-49) adults. The study is broken down into four treatment groups. Each group will enroll 100 subjects, for a total of 400 subjects. Groups A-C will receive one of three dose levels of the Quadrivalent VLP vaccine, and Group D will receive a commercially available trivalent influenza vaccine (TIV). The study will also evaluate the safety and tolerability of the Quadrivalent VLP vaccine formulations.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female, 18-49 years of age
2. Willing and able to give informed consent prior to study enrollment
3. Able to comply with study requirements
4. Women of child-bearing potential must have a negative urine pregnancy test at vaccination, will be advised through the Informed Consent process to avoid becoming pregnant over the duration of the study, and must assert that they will employ an effective form of birth control for the duration of the study. Acceptable forms of birth control are: credible history of continuous abstinence from heterosexual activity, or prior surgical sterilization, hormonal contraceptives (oral, injectable, implant, patch, ring), barrier contraceptives (condom or diaphragm), and intrauterine device (IUD). Women with an adequately documented history of surgical sterility are exempt from urine pregnancy testing.

Exclusion Criteria:

1. Any ongoing, symptomatic acute or chronic illness requiring medical or surgical care.

   * Asymptomatic conditions or findings (e.g., mild hypertension, dyslipidemia) that are not associated with evidence of end-organ damage are not exclusionary provided that they are being appropriately managed and are clinically stable (i.e., unlikely to result in symptomatic illness within the time-course of this study) in the opinion of the investigator.
   * Acute or chronic illnesses or conditions which may be reasonably predicted to become symptomatic if treatment were withdrawn or interrupted are exclusionary, even if stable.
   * Acute or chronic illnesses reasonably expected to be associated with increased risks associated with influenza (e.g., cardio-pulmonary diseases, diabetes mellitus, renal or hepatic dysfunction, hemoglobinopathies) are exclusionary, even if stable.
   * Note that illnesses or conditions may be exclusionary, even if otherwise stable, due to therapies used to treat them (see exclusion criteria 2,5,8,9).
2. Participation in research involving investigational product (drug/ biologic/ device) within 45 days before planned date of first vaccination
3. History of a serious reaction to prior influenza vaccination, known allergy to constituents of licensed TIV (e.g., egg proteins) or polysorbate-80.
4. History of Guillain-Barré Syndrome (GBS) within 6 weeks following a previous influenza vaccine.
5. Received any vaccine in the 4 weeks preceding the study vaccination and any influenza vaccine within six months preceding the study vaccination.
6. History of receipt of any avian influenza vaccine containing an H5 antigen, or known exposure to birds infected with an H5 virus.
7. Any known or suspected immunosuppressive illness, congenital or acquired, based on medical history and/or physical examination.
8. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccine. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose greater or equal to 10mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted.
9. Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or during the study.
10. Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature >38.0°C on the planned day of vaccine administration.
11. Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled or could interfere with evaluation of the vaccine or interpretation of study results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).
12. Known disturbance of coagulation.
13. Women who are breastfeeding or plan to become pregnant during the study.
14. Suspicion or recent history (within one year of planned vaccination) of alcohol or other substance abuse.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of the quadrivalent VLP vaccine using HAI responses. | Up to 6 months
  Derived/calculated endpoints based on:
  Seroconversion rate (SCR) Seroprotection rate (SPR) Geometric mean titer (GMT) Geometric mean ratio (GMR)
Safety of three quadrivalent VLP vaccine formulations. adverse events, Medically Attended Events (MAEs), Serious Adverse Events (SAEs), and Significant New medical Conditions (SNMCs) | Up to 6 months
  Number and percentage of subjects with solicited local and systemic adverse events over the seven days post-injections; all adverse events (including adverse changes in clinical laboratory parameters) over 21 days post-injections; and Medically Attended Events (MAEs), Serious Adverse Events (SAEs), and Significant New medical Conditions (SNMCs) through six months.

SECONDARY OUTCOMES:
Immunogenicity of each quadrivalent VLP vaccine formulation measured by neuraminidase inhibition (NAI) | Up to 6 months
  Derived/calculated endpoints based on:
  Two fold and four fold increases in NAI titer Geometric mean titer (GMT) Geometric mean ratio (GMR)

CONTACTS AND LOCATIONS:
Overall Officials: D Nigel Thomas, Ph.D., Study Director — Novavax
Locations (5):
- United States (5):
  - Anaheim Clinical Trials, Anaheim, California
  - Miami Research Associates, Miami, Florida
  - Johnson County Clin Trials, Lenexa, Kansas
  - Meridian Clinical Research, Omaha, Nebraska
  - Clinical Trials of Texas, San Antonio, Texas

REFERENCES:
- See also: Novavax, Inc. — http://www.novavax.com